CLINICAL TRIAL: NCT06021912
Title: Evaluating the Efficacy of Allergen Immunotherapy in the Management of Allergic Asthma and Rhinitis
Brief Title: e-ITAG Allergen Immunotherapy in the Management of Allergic Asthma
Acronym: EITAG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: General Administration of Military Health, Tunisia (Network)
Responsible Party: Principal Investigator, Hedi Gharsallah, DR SELSABIL Daboussi, General Administration of Military Health, Tunisia
Other Study IDs: efficacity of EITAG
Record Dates: First submitted 2023-08-26; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Study the Efficacy of ITA in Patients With Allergic Asthma or Allergic Rhinitis or Allergic Rhinitis Compared With Conventional Treatment
Keywords: ITA ASTHMA ALLERGIC RHINITIS
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ITA GROUP: Patients with asthma or allergic rhinitis who have received allergen immunotherapy (ITA).
  Interventions: Drug: Immunotherapy
- STANDARD TREATMENT: patients with asthma or allergic rhinitis who have received standard allergen treatment.
  Interventions: Drug: Immunotherapy

INTERVENTIONS:
Drug: Immunotherapy — Sublingual immunotherapy

SUMMARY:
Allergy is defined as a specific abnormal and excessive reaction of the immune system to exposed allergen .

This reaction is reproducible with each new exposure allergen . A recent study by The European Academy of Allergy and Clinical Immunology" (EAACI) estimates that 30% of the population suffers from allergic rhinitis and/or conjunctivitis, 20% of children suffer from asthma, and 8% of the population suffers from food allergies in Europe, with a clear increase in prevalence.

Allergenic immunotherapy (AIT) remains a corner stone in the treatment of allergic diseases. It involves administering an increasing dose of allergens to induce immunological tolerance. The efficacy and safety of ITA have already been demonstrated. However, patient response is highly heterogeneous. This findinf illustrates the value of biomarkers in the selection of patients, enabling prediction of response to ITA and follow-up.

DETAILED DESCRIPTION:
This is a prospective, observationel study conducted in Pneumology Department at the Military Hospital in collaboration with the Immunology Laboratory

We followed patients in 2 groups:

Group 1: patients with asthma or allergic rhinitis who had received allergen immunotherapy (AIT). Group 2: patients with asthma or allergic rhinitis who received a conventional treatment

ELIGIBILITY:
Inclusion Criteria Patients with symptoms of Asthma or moderate or severe persistent allergic rhinitis allergic rhinitis, with a positive prick test or specific IgE assay demonstrating the presence of allergens (1 or 2 allergens). A significant impact on the patient's quality of life Rhinitis associated with tracheitis or mild-to-moderate asthma. Patients with poorly controlled asthma despite optimal treatment Ineffective drug treatment Patients willing to adhere to our research protocol

Exclusion Criteria:

Patients with multi-allergenic asthma (more than 2 allergens) Pregnancy (at the time of ITA initiation). Autoimmune disease Immunosuppressive treatment Poorly controlled asthma HIV infection Cancer Severe psychiatric disorders. Cardiovascular diseases with a risk of complications during administration of adrenaline. Use of beta-blockers. Treatment with ACE inhibitors. Persistent lesions of the oral mucosa (chronic oral aphthosis periodontitis, etc.). Worsening of rhinitis. Acute febrile state. Recent administration of another vaccine (in this case, the ITA should not be administered on the same day).

ITA should not be administered on the same day).

Ages: 5 Years to 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with symptoms of Asthma or moderate or severe persistent allergic rhinitis allergic rhinitis, with a positive prick test or specific IgE
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Increase in IGG1, IGG4 | After 6 month of ITA
  increase in IGG1, IGG4 after ITA treatment compared to conventional treatment group (prik test /ratio of IGE/IG4/ rate of significant increase is > 25%.
Deacresed basophil activation | After 6 month of ITA
  activation of basophils by the presence of the CD203c marker in the ITA group compared with the conventional treatment group

SECONDARY OUTCOMES:
Evalution AQLQS score(QUALITY OFLIFE) | After 6 month of ITA
  Assessing the quality of life in asthma patient by AQLQS score/ ACQ/ ARIA

CONTACTS AND LOCATIONS:
Overall Officials: SELSABIL DABOUSSI, MD, Principal Investigator — Pneumologie
Locations (1):
- Military Hospital of Tunis, Tunis, Montfleury, Tunisia

IPD SHARING:
Plan to Share IPD: No